CLINICAL TRIAL: NCT05730049
Title: Assessing the Efficacy of Transcutaneous Auricular Vagus Nerve Stimulation as an Anti-inflammatory Treatment Following Spinal Cord Injury
Brief Title: Neuromodulation as an Anti-inflammatory Treatment in SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12901
Record Dates: First submitted 2023-01-13; First posted 2023-02-15 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Inflammation
Keywords: Vagus Nerve Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Inflammation

STUDY DESIGN:
Intervention Model Description: Eligible participants who consent to study participation will be randomized to one of two groups: active taVNS, or sham taVNS. Each group will undergo 1 hour of the respective treatment.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active taVNS (Experimental): Stimulation will target the auricular branch of the vagus nerve by applying stimulation to the cymba conchae region of the ear using the NEMOS® taVNS device (taVNS Technologies, Erlangen, Germany). To achieve adequate stimulation while avoiding unpleasant or painful sensations, the stimulation intensity will be gradually increased in increments of 0.1mA until the subjective pain threshold is reached, and then reduced to a stimulus intensity just below the individuals pain threshold (expected range based on prior studies 1 - 3.2mA. Pulse width will be set at 100μs and frequency will be set at 25Hz as performed in a previous protocol in stroke patients. Stimulation will be applied for a duration of 1 hour.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation
- Sham taVNS (Sham Comparator): The control group will receive the same stimulation parameters but will have the earpiece placed in the sham position such that stimulation is applied to the earlobe and does not activate the vagus nerve.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — Stimulation will target the auricular branch of the vagus nerve by applying stimulation to the cymba conchae region of the ear using the NEMOS® taVNS device (taVNS Technologies, Erlangen, Germany). To achieve adequate stimulation while avoiding unpleasant or painful sensations, the stimulation intensity will be gradually increased in increments of 0.1mA until the subjective pain threshold is reached, and then reduced to a stimulus intensity just below the individuals pain threshold (expected range based on prior studies 1 - 3.2mA(3). Pulse width will be set at 100μs and frequency will be set at 25Hz as performed in a previous protocol in stroke patients(3). The control group will receive the same stimulation parameters but will have the earpiece placed in the sham position such that stimulation is applied to the earlobe and does not activate the vagus nerve(4).
  Other Names: NEMOS® taVNS device

SUMMARY:
The goal of this single-blinded randomized, controlled trial is to assess the impact of 1-hour of active transcutaneous auricular vagus nerve stimulation (taVNS) vs sham taVNS on serum biomarkers of the inflammatory reflex and inflammation in individuals with spinal cord injury.

The main question it aims to answer is: whether taVNS is a safe and effective anti-inflammatory intervention for individuals with SCI. Participants will perform a single 1-hour bout of the respective taVNS treatment with blood draws prior to treatment, immediately following treatment, and 24 hours following treatment. Changes in biomarkers between the active and sham taVNS conditions will be compared.

DETAILED DESCRIPTION:
Chronic inflammation is very common among individuals living with spinal cord injury (SCI) and contributes to a number of health complications(1). Drug treatments are available to help reduce inflammation, however, many patients are unresponsive, become resistant or experience adverse effects such as increased risk of infection(2). There is a need for other treatments which reduce inflammation while avoiding harmful side effects.

It is now understood that the nervous systems plays an important role in regulating the immune system and controlling inflammation. The vagus nerve has been shown to be a particularly important part of the nervous system in terms of limiting inflammation. However, SCI causes disruption to the nervous system, including reduced activity of the vagus nerve. This may contribute to excessive inflammation. New technologies have been developed that allow the vagus nerve to be activated by electrically stimulating a part of the ear. This technique called vagus nerve stimulation (VNS) has been shown to help reduce inflammation in numerous populations. However, it has not been assessed in individuals with SCI. This study will assess if stimulating the vagus nerve can be a safe and effective way to reduce inflammation in individuals with SCI.

To assess this, 30 individuals with SCI who agree to participate will be randomly assigned to receive either active VNS treatment or sham treatment (whereby the device will placed in such a way that it does not stimulate the vagus nerve). Participants will not be aware of which group they are in. The study will take place over a 2-day period. On day one, participants will arrive in the morning for a fasted blood draw to assess baseline inflammation. Following the blood draw, participants will receive 1-hour of either the active or sham VNS therapy. Immediately following VNS therapy a second blood draw will be performed. On day 2 participants will be asked to return at the same time of day to complete a final fasted blood draw. This will allow for the assessment of how well the therapy activated 2 key anti-inflammatory pathways controlled by the vagus nerve and resulting changes in inflammation (immediate and 24-hour post).

It is expected that VNS therapy will be well-tolerated, safe and effective at reducing inflammation in individuals with SCI. If this is shown, VNS may prove to be a simple and cost-effective means of reducing chronic inflammation in individuals with SCI and may help to replace and/or reduce the need for other pharmaceutical drugs which are associated with adverse health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any level of severity of spinal cord injury
* 18 years of age or older

Exclusion Criteria:

* pregnant or attempting to become pregnant
* people with active implants (e.g. cochlear implant, implanted vagus nerve stimulator, cardiac pacemaker)
* people with cerebral shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Biomarkers Immediately Following Intervention | Baseline - Immediately Following Intervention
  Change in serum concentrations of the pro-inflammatory cytokines tumour necrosis factor-alpha (TNF-alpha), C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and interferon-gamma (IFN-y) immediately following intervention. Change in serum concentrations of acetylcholine immediately following intervention will be assessed as an indicator of the activity of the cholinergic anti-inflammatory pathway, and the change in cortisol immediately following intervention will be assessed as an indicator of the activity of the neuro-endo-immune pathway.
Change in Serum Biomarkers 24-hours Following Intervention | Baseline - 24-hour Post Intervention
  Change in serum concentrations of the pro-inflammatory cytokines tumour necrosis factor-alpha (TNF-alpha), C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and interferon-gamma (IFN-y) 24-hours following intervention. Change in serum concentrations of acetylcholine 24-hours following intervention will be assessed as an indicator of the activity of the cholinergic anti-inflammatory pathway, and the change in cortisol 24-hours following intervention will be assessed as an indicator of the activity of the neuro-endo-immune pathway.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events During or Immediately Following Intervention | Immediately Following Intervention
  All adverse events which occur during or immediately following the intervention will be recorded during the study visit and compared between the taVNS and sham conditions. A description of the adverse event, number of events, and total number of participants affected will be recorded.
Incidence of Treatment-Emergent Adverse Events 24-hours Following Intervention | 24-hour Post intervention
  All adverse events which occur within 24-hours following the intervention will be self-reported by participants and recorded and compared between the taVNS and sham conditions. A description of the adverse event, number of events, and total number of participants affected will be recorded.
Time required to recruit 30 participants | Immediately following 6-month recruitment period
  The success of participant recruitment will be assessed based on the time required to recruit the target 30 participants. Completion of recruitment in under 6-months will be considered successful.
Program Completion Rates | Immediately after intervention
  Program completion rates will be assessed by the number of participants who completed the entire 1-hour intervention in its entirety.
Participant Satisfaction with Intervention | 24-hour Post intervention
  Participant satisfaction with the intervention will be assessed via an 11-point visual analog scale (VAS) with scores ranging from 0-10 whereby 0 reflects complete dissatisfaction and 10 reflects complete satisfaction as well as qualitatively via participant feedback.

CONTACTS AND LOCATIONS:
Overall Officials: David J. Allison, PhD., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, St Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison DJ, Ditor DS. The common inflammatory etiology of depression and cognitive impairment: a therapeutic target. J Neuroinflammation. 2014 Sep 2;11:151. doi: 10.1186/s12974-014-0151-1. PMID 25178630
- [Background] Tynan A, Brines M, Chavan SS. Control of inflammation using non-invasive neuromodulation: past, present and promise. Int Immunol. 2022 Jan 22;34(2):119-128. doi: 10.1093/intimm/dxab073. PMID 34558623
- [Background] Redgrave JN, Moore L, Oyekunle T, Ebrahim M, Falidas K, Snowdon N, Ali A, Majid A. Transcutaneous Auricular Vagus Nerve Stimulation with Concurrent Upper Limb Repetitive Task Practice for Poststroke Motor Recovery: A Pilot Study. J Stroke Cerebrovasc Dis. 2018 Jul;27(7):1998-2005. doi: 10.1016/j.jstrokecerebrovasdis.2018.02.056. Epub 2018 Mar 23. PMID 29580658
- [Background] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069